CLINICAL TRIAL: NCT04776252
Title: A Phase 3 Open-label Rollover Clinical Study of Doravirine/Islatravir (DOR/ISL) Once-daily for the Treatment of HIV-1 Infection in Participants Who Previously Received DOR/ISL in a Phase 2 or Phase 3 DOR/ISL Clinical Study
Brief Title: Open-label, Follow-up of Doravirine/Islatravir (DOR/ISL 100 mg/0.75mg) for Participants With Human Immunodeficiency Virus-1 (HIV-1) Infection (MK-8591A-033)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8591A-033; MK-8591A-033 (Other: MSD); jRCT2031210528 (Registry Identifier: jRCT); 2024-512215-53-00 (Registry Identifier: EU CT); U1111-1304-7926 (Registry Identifier: UTN); 2020-001191-14 (EudraCT Number)
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-8591A (Experimental): Fixed dose combination (FDC) tablet of 100 mg doravirine, 0.75 mg islatravir taken orally, once daily for up to 192 weeks.
  Interventions: Drug: MK-8591A

INTERVENTIONS:
Drug: MK-8591A — FDC tablet of 100 mg doravirine, 0.75 mg islatravir taken orally, once daily for up to 192 weeks

SUMMARY:
The safety and tolerability of MK-8591A, a 2-drug fixed dose combination (FDC) of doravirine (100mg) and islatravir (0.75mg) [DOR/ISL 100 mg/0.75 mg) will be evaluated in participants with Human Immunodeficiency Virus -1 (HIV-1) who were treated with DOR and ISL in earlier clinical studies.

DETAILED DESCRIPTION:
As of Amendment 12, participants will have the option to continue receiving DOR/ISL (100 mg/0.75 mg) until treatment alternatives are identified, or up to Week 288 given that participants are still deriving benefit, based on individual benefit/risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* Is currently receiving DOR 100 mg/ISL 0.75 mg adult FDC tablet in an MSD-sponsored clinical study and has completed the last treatment visit.
* Is considered by the investigator to have derived clinical benefit from receiving DOR/ISL and for whom further treatment with DOR/ISL is considered clinically appropriate.
* Female is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP); or is a non-pregnant WOCBP who agrees to the following during the intervention period and for at least 6 weeks after the last dose of study intervention: Not be sexually active, or if sexually active, to use an acceptable method of contraception; or is pregnant and continues to receive study intervention (where allowed by local regulations and as appropriate based on available data/local standard-of-care guidelines)

Exclusion Criteria:

* Is taking or is anticipated to require any prohibited therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2029-05-29 (Estimated); Study Completion 2029-05-29 (Estimated)

PRIMARY OUTCOMES:
Participants with serious adverse events (SAEs) | Up to Week 198
  Percentage of participants with serious adverse events (SAEs)
Participants who discontinued due to an adverse event (AE) | Up to Week 192
  Percentage of participants who discontinued study treatment due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (93):
- United States (18):
  - Pueblo Family Physicians ( Site 0010), Phoenix, Arizona
  - One Community Health ( Site 0045), Sacramento, California
  - Whitman-Walker Institute ( Site 0039), Washington D.C., District of Columbia
  - Georgetown University Medical Center-Clinical Trials Unit Division of Infectious Diseases ( Site 002, Washington D.C., District of Columbia
  - Midway Immunology and Research Center ( Site 0033), Ft. Pierce, Florida
  - Orlando Immunology Center ( Site 0017), Orlando, Florida
  - Bliss Healthcare Services-Research ( Site 0030), Orlando, Florida
  - Triple O Research Institute, P.A ( Site 0031), West Palm Beach, Florida
  - Chatham County Health Department - Chatham CARE Center-Infectious Disease ( Site 0015), Savannah, Georgia
  - Northstar Healthcare ( Site 0003), Chicago, Illinois
  - KC CARE Health Center-Clinical Trials ( Site 0012), Kansas City, Missouri
  - ID Care ( Site 0028), Hillsborough, New Jersey
  - Icahn School of Medicine at Mount Sinai-Clinical and Translational Research Center ( Site 0006), New York, New York
  - Penn Medicine: University of Pennsylvania Health System-Perelman Center for Advanced Medicine ( Site, Philadelphia, Pennsylvania
  - St Hope Foundation ( Site 0041), Bellaire, Texas
  - North Texas Infectious Diseases Consultants, P.A-Research ( Site 0004), Dallas, Texas
  - Texas Center for Infectious Disease Associates-Clinical Research ( Site 0026), Fort Worth, Texas
  - The Crofoot Research Center ( Site 0008), Houston, Texas
- Australia (3):
  - Holdsworth House Medical Practice ( Site 0700), Darlinghurst, New South Wales
  - St Vincent's Hospital-IBAC ( Site 0702), Sydney, New South Wales
  - Fiona Stanley Hospital ( Site 0706), Murdock, Western Australia
- Canada (7):
  - Sheldon M. Chumir Health Centre-Southern Alberta Clinic ( Site 0106), Calgary, Alberta
  - Vancouver Infectious Diseases Centre ( Site 0100), Vancouver, British Columbia
  - Hamilton Health Sciences- Urgent Care Centre-SIS Clinic ( Site 0109), Hamilton, Ontario
  - Maple Leaf Research ( Site 0105), Toronto, Ontario
  - Toronto General Hospital ( Site 0104), Toronto, Ontario
  - Clinique de médecine Urbaine du Quartier Latin ( Site 0110), Montreal, Quebec
  - Clinique Medicale lActuel ( Site 0108), Montreal, Quebec
- Chile (4):
  - Biomedica Research Group-Infectology ( Site 0201), Santiago, Region M. de Santiago
  - Centro de Investigacion Clinicadela Universidad Catolica ( Site 0204), Santiago, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile ( Site 0200), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco-Unidad de Investigación Clínica ( Site 0202), Temuco, Región de la Araucanía
- Fundacion Valle del Lili- CIC ( Site 0300), Cali, Valle del Cauca Department, Colombia
- France (13):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 1504), Nice, Alpes-Maritimes
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 1516), Dijon, Bourgogne-Franche-Comté
  - CHU de Bordeaux Hop St ANDRE-Médecine interne et maladies infectieuses ( Site 1512), Bordeaux, Gironde
  - CHU de Toulouse-Infectious Disease-Tropical Diseases ( Site 1505), Toulouse, Haute-Garonne
  - CHU Charles Nicolle-Inefectious disease ( Site 1506), Rouen, Haute-Normandie
  - Hospital La Colombière ( Site 1518), Montpellier, Herault
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu ( Site 1517), Nantes, Loire-Atlantique
  - Tourcoing Hospital-Service Universitaire des Maladies Infectieuses et du Voyageur ( Site 1519), Tourcoing, Nord
  - Hôpital de la Croix Rousse-Service des Maladies infectieuses et tropicales ( Site 1503), Lyon, Rhone
  - Hôpital Bichat - Claude-Bernard-infectious diseases ( Site 1523), Paris
  - Hôpital Avicenne ( Site 1502), Bobigny, Île-de-France Region
  - Hôpital Saint-Louis-Infectious Diseases and tropical diseases ( Site 1511), Paris, Île-de-France Region
  - Pitie Salpetriere University Hospital-Infectious Disease - Tropical Diseases ( Site 1508), Paris, Île-de-France Region
- Medizinische Hochschule Hannover-Department of Immunology and Rheumatology ( Site 1661), Hanover, Lower Saxony, Germany
- Italy (4):
  - Fondazione Policlinico Universitario Agostino Gemelli-UOC Malattie Infettive ( Site 1606), Rome, Lazio
  - Ospedale San Raffaele-U.O. Malattie Infettive ( Site 1602), Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo-Dipartimento di Malattie Infettive: SC Malattie Infettive (, Pavia, Lombardy
  - Ospedale Luigi Sacco-UOC Malattie Infettive I ( Site 1600), Milan, Milano
- Japan (5):
  - National Hospital Organization Nagoya Medical Center ( Site 0903), Nagoya, Aichi-ken
  - Tokyo Medical University Hospital ( Site 0904), Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine ( Site 0901), Shinjyuku-ku, Tokyo
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research ( Site 09, Osaka
  - Tokyo Metropolitan Komagome Hospital ( Site 0906), Tokyo
- Christchurch Hospital-Infectious Diseases ( Site 0800), Christchurch, Canterbury, New Zealand
- Poland (4):
  - Wrocl.Centr.Zdrowia SPZOZ Osr. Prof-Lecz Ch. Zak. i Terapii Uzaleznien ( Site 1703), Wroclaw, Lower Silesian Voivodeship
  - EMC Instytut Medyczny S. A. Przychodnia przy ul. Lowieckiej we Wroclawiu ( Site 1700), Wroclaw, Lower Silesian Voivodeship
  - Wojewódzki Szpital Zakaźny w Warszawie ( Site 1702), Warsaw, Masovian Voivodeship
  - WSS im. W Bieganskiego O. Chorob Zakaznych i Hepatologii-F ( Site 1701), Ód, Łódź Voivodeship
- Russia (8):
  - Kuzbasskiy Center for the Prevention and Control of AIDS ( Site 2305), Kemerovo, Kemerovo Oblast
  - Krasnoyarsk Regional Center for the Prevention and Control of AIDS ( Site 2304), Krasnoyarsk, Krasnoyarsk Krai
  - Republican Clinical Infectious Hospital ( Site 2300), Saint Petersburg, Leningradskaya Oblast'
  - Moscow Infectious Diseases Clinical Hospital Number 2 ( Site 2306), Moscow, Moscow
  - Scientific Advisory Clinical Diagnostic Center Central Resea-Federal AIDS Center ( Site 2302), Moscow, Moscow
  - Saint-Petersburg Center for Prophylactic of AIDS and Infecti-Saint-Petersburg Center for Prophylact, Saint Petersburg, Sankt-Peterburg
  - Smolensk Center for prevention and control of AIDS ( Site 2308), Smolensk, Smolensk Oblast
  - Republican Clinical Hospital for Infectious Diseases A.F. Agafonova ( Site 2303), Kazan', Tatarstan, Respublika
- South Africa (6):
  - Josha Research ( Site 2403), Bloemfontein, Free State
  - Ezintsha ( Site 2404), Johannesburg, Gauteng
  - Mediclinc Muelmed ( Site 2401), Pretoria, Gauteng
  - King Edward VIII Hospital ( Site 2410), Durban, KwaZulu-Natal
  - Wentworth Hospital ( Site 2400), Durban, KwaZulu-Natal
  - Desmond Tutu Health Foundation ( Site 2402), Cape Town, Western Cape
- Spain (7):
  - Hospital General Universitario de Elche-Infectius Disease ( Site 1908), Elche, Alicante
  - Hospital Germans Trias i Pujol-Fundació Lluita contra la Sida ( Site 1901), Badalona, Barcelona
  - HOSPITAL CLÍNIC DE BARCELONA-Infection Day Hospital ( Site 1900), Barcelona, Catalonia
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-Unidad de Enfermedades Infecciosas ( Site 1903), Madrid, Madrid, Comunidad de
  - Hospital Universitario Infanta Leonor ( Site 1906), Madrid
  - Hospital Universitario Fundación Jiménez Díaz-Internal Medicine. Infectious disease ( Site 1902), Madrid
  - Hospital Universitario La Paz-Internal Medicine ( Site 1904), Madrid
- Switzerland (6):
  - University Hospital Basel-Infectiology ( Site 2002), Basel, Canton of Aargau
  - Hôpitaux Universitaires de Genève (HUG)-Infectious Disease Department ( Site 2004), Geneva, Canton of Geneva
  - Cantonal Hospital St.Gallen ( Site 2001), Sankt Gallen, Canton of St. Gallen
  - UniversitätsSpital Zürich ( Site 2000), Zurich, Canton of Zurich
  - Ospedale Regionale di Lugano, Sede Civico-Servizio Malattie Infettive ( Site 2005), Lugano, Canton Ticino
  - Inselspital Bern-Inselspital Infektiologie ( Site 2003), Bern
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust ( Site 2104), East Sussex, Brighton And Hove
  - Southmead Hospital ( Site 2103), Bristol, Bristol, City of
  - Royal Free Hospital ( Site 2102), London, England
  - King's College Hospital ( Site 2101), London, England
  - North Manchester General Hospital ( Site 2105), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26182&tenant=MT_MSD_9011